CLINICAL TRIAL: NCT02734693
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of Dasotraline in Children Aged 6 to 12 Years With Attention-Deficit Hyperactivity Disorder (ADHD) in a Laboratory Classroom Setting
Brief Title: A Study to Evaluate the Efficacy and Safety of Dasotraline in Children 6 to 12 Years of Age With Attention-Deficit Hyperactivity Disorder (ADHD) in a Simulated Classroom Setting.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEP360-305
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Attention-Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention-Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine; SEP 225289

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasotraline 4mg (Experimental): Dasotraline capsule 4mg/day
  Interventions: Drug: dasotraline 4mg
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: dasotraline 4mg — dasotraline 4mg/day
  Other Names: SEP-225289
  Arms: Dasotraline 4mg
Other: Placebo — placebo/day
  Other Names: Placebo comparitor
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and safety of dasotraline in children 6 years of age to 12 years of age with Attention-Deficit Hyperactivity Disorder (ADHD) in a simulated classroom setting.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, efficacy and safety study in children with ADHD in a laboratory classroom setting. The study will be comprised of 3 periods: Screening (up to 35 days) including a 3 - 5 day ADHD medication washout prior to Day -1; Double-blind randomized treatment with either dasotraline (4 mg/day) or placebo for14 days; and End of Study (EOS) Visit (7 days after last dose). Prior to the start of treatment (Day 1) and following the conclusion of the double-blind period (Day 15), subjects will undergo a full-day laboratory classroom evaluation during which approximately 12 to 18 subjects will be assessed. Each laboratory classroom day will include seven 30-minute simulated classroom sessions where trained observers will assess subjects using the Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Scale. In addition during each classroom session, a 10-minute math test (Permanent Product Measure of Performance [PERMP]) will be administered to evaluate sustained attention and effort. Seven (± 2) days after the last dose of study drug, subjects will return to the clinic and complete safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is 6 - 12 years old, inclusive at screening and randomization. 2. At least one of the subject's parents/legal guardians must give written informed consent, including privacy authorization, prior to study participation. The subject will provide informed assent prior to study participation.

  3. Subject meets Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined presentation) at screening established by a comprehensive psychiatric evaluation that reviews DSM-5 criteria and confirmed using the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (K-SADS-PL) at screening.

  4. Subject is currently on a treatment regimen of a methylphenidate formulation within the approved labeled dose range for ADHD for at least 6 weeks prior to Day -7 with the same dose level for at least 1 week immediately prior to Day -7. Note: if any doses of methylphenidate were missed during the week prior to Day-7, the subject's eligibility will be discussed with the Medical Monitor.

  5. In the opinion of the investigator, methylphenidate well tolerated and clinically effective based on clinical assessment and informant interview, as well as, review of available medical records. Note: The ADHD Rating Scale Version IV - Home Version (modified for investigator administration) (ADHD-RS-IV HV) will be administered at Screening by the investigator to inform clinical evaluation.

  6. Subject is male or a non-pregnant, non-lactating female. 7. Subject, if female, must not be pregnant or breastfeeding, and if ≥ 8 years of age must have a negative serum pregnancy test at screening.

  8. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must practice true abstinence (consistent with lifestyle) and must agree to remain abstinent or agree to use an effective and medically acceptable form of birth control, from the time of informed consent/assent to at least 14 days after the last dose of the study drug has been taken.

  9. Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical and neurological examinations, medical history, and clinical laboratory values (hematology, chemistry, and urinalysis). Note: If any of the hematology, chemistry, or urinalysis results are not within the laboratory's reference range, then the subject can be included only if the investigator determines the deviations to be not clinically relevant.

  10. Subject is within the 3rd to 97th percentile for gender specific body mass index (BMI)-for-age from the World Health Organization (WHO) growth charts and weighs at least 21 kg.

  11. Subject must report a history of being able to swallow capsules. 12. Subject and subject's parent/legal guardian must be able to fully comprehend the informed consent/assent forms, understand and be willing and able to comply with all study procedures and visit schedule, and be able to communicate satisfactorily with the investigator and study coordinator.

Exclusion Criteria:

* 1. Subject or parent/legal guardian has commitments during the study that would interfere with attending study visits.

  2. Subject, on Day 1, has not demonstrated evidence of worsening of ADHD symptoms as measured by ADHD-RS-IV HV total score ≥ 26 and at least a 30% worsening in ADHD-RS-IV HV total score since the last assessment and following a minimum 72-hour washout from prior methylphenidate treatment.

  3. Subject is currently being treated for ADHD with an amphetamine-based product, or has been treated with an amphetamine-based product in the 6 weeks prior to the start of screening.

  4. Subject is currently being treated for ADHD with a non-methylphenidate product, or has been treated with a non-methylphenidate product in the 6 weeks prior to the start of screening.

  5. Subject has failed 2 adequate courses (dose and duration) of stimulant or non-stimulant treatment for ADHD, as judged by the investigator.

  6. Subject currently has a diagnosis of asthma that has required daily treatment with bronchodilators or nebulizer treatments in the 30 days prior to screening and/or who may require daily treatments with these agents over the course of the trial. Intermittent use of bronchodilators is not exclusionary. Subjects who have a history of requiring persistent asthma treatment should be discussed with the medical monitor prior to randomization.

  7. Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition (eg, malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion. Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the medical monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if controlled) must be discussed with the medical monitor during screening.

  8. Subject has a history or presence of abnormal ECGs, which in the investigator's opinion is clinically significant. Screening site ECGs will be centrally over-read, and eligibility will be determined by the investigator based on the results of the over-read report.

  9. Subject has any diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, any history of psychosis, autism spectrum disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances. Note: Subjects with oppositional defiant disorder (ODD) are permitted to enroll in the study as long as ODD is not the primary focus of treatment.

  10. Subject has generalized anxiety disorder or panic disorder that has been the primary focus of treatment at any time during the 12 months prior to screening or that has required pharmacotherapy any time during the 6 months prior to screening.

  11. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood (eg, Duchenne Muscular dystrophy, myasthenia gravis, or other neurologic or serious neuromuscular disorders), or history of persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, drug-induced seizure, or alcohol withdrawal seizure is exclusionary. Subject taking anticonvulsants for seizure control currently or within the past 2 years is not eligible for study participation.

  12. Subject has uncontrolled thyroid disorder as evidenced by thyroid stimulating hormone (TSH) ≤ 0.8 x the lower limit of normal (LLN) or ≥ 1.25 x the upper limit of normal (ULN) for the reference laboratory.

  13. Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for any lifetime history on the C-SSRS Children's Lifetime/Recent assessment at screening.

  14. Subject has any history of attempted suicide or clinically significant suicidal ideation, in the opinion of the investigator.

  15. Subject has a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions or has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulations.

  16. Subject has history of intolerance (safety) or lack of efficacy to stimulants.

  17. Subject has taken any antipsychotic medication within 6 months prior to screening.

  18. Subject has taken any herbal and/or complementary treatments, eg, St. John's Wort, within 7 days prior to Day 1.

  19. Subject has taken any antidepressant medication (eg, bupropion, selective serotonin reuptake inhibitor [SSRI]/ serotonin norepinephrine reuptake inhibitor [SNRI], tricyclic, etc) within 7 days prior to Day 1.

  20. Subject has taken any monoamine oxidase [MAO] inhibitor within 21 days prior to Day 1.

  21. Subject is currently undergoing Cognitive Behavioral Therapy (CBT) for the treatment of ADHD, has initiated behavioral therapy (including school based interventions) less than 1 month prior to screening, or is receiving behavioral therapy and in the opinion of the investigator will not be able to follow a stable routine for the duration of the study. Note: Unavoidable changes in school-based interventions that occur during study participation will not be exclusionary, but should be documented by the investigator, to the extent possible.

  22. Subject or subject's family anticipates a move outside the geographic range of investigative site during the study period, or plans extended travel inconsistent with the recommended visit interval during study duration.

  23. Subject has history of, or current malignancy except for non-melanomatous skin cancer.

  24. Subject has history of positive test for Hepatitis B surface antigen or Hepatitis C antibody.

  25. Subject is known to have tested positive for human immunodeficiency virus (HIV).

  26. Subject has participated in a classroom study within 6 months prior to the start of screening or has participated in any other clinical study with an investigational drug/product within 90 days prior to the start of screening or is currently participating in another clinical trial.

  27. Subject shows evidence of substance or alcohol use or is currently using tobacco or other nicotine-containing products, or has a positive urine drug screen (UDS) at screening. Note: Subjects with a positive UDS may be allowed to continue in the study, provided that the investigator determines that the positive test is as a result of taking medications as prescribed after consultation with the medical monitor.

  28. Subject is taking any disallowed medications for chronic treatment. 29. Subject has previously been enrolled in a clinical trial of dasotraline (SEP-225289).

  30. Subject's parent/legal guardian is an investigational site staff member or the relative of an investigational site staff member.

  31. Subject is, in the opinion of the investigator, unsuitable in any other way to participate in this study.

  32. Subject's sibling or family member living in the same household is participating in the same laboratory classroom cohort for this study.

  33. Subject is unable to perform at the basic level of the standardized math test as defined in the laboratory classroom manual.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sunovion Pharamceuticals Inc.
Locations (5):
- United States (5):
  - Avida Inc, Newport Beach, California
  - Meridien Research, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Ltd, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasotraline 6mg: Dasotraline capsule 6mg/day
Period: Overall Study
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Started | 56 | 56 | 20
Completed | 50 | 53 | 17
Not Completed | 6 | 3 | 3
Not completed — Adverse Event | 1 | 3 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg | Total
Number analyzed (Participants) | 56 | 56 | 20 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 56 | 20 | 132
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (1.86) | 9.3 (1.76) | 9.9 (1.69) | 9.6 (1.8)
Age, Customized [Number; unit: participants]
  6-9 years | 24 | 30 | 7 | 61
  10-12 years | 32 | 26 | 13 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 6 | 41
  Male | 38 | 39 | 14 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 19 | 5 | 35
  Not Hispanic or Latino | 45 | 37 | 15 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 23 | 25 | 6 | 54
  White | 31 | 26 | 13 | 70
  More than one race | 1 | 3 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 20 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Day 15 in , ADHD Symptoms as Measured by Mean Swanson,Kotkin,Agler,M-Flynn, Pelham Rating Scale(SKAMP)-Combined Score Obtained From an Average of the 7 Assessments Collected Across the 12-hour Classroom Day(12 to 24 Hours Postdose)
Description: The Swanson, Kotkin, Agler, M-Flynn, Pelham Rating Scale (SKAMP) scale is a 13-item independent observer rating of subject impairment of classroom observed behaviors. Each item is rated on a 7-point impairment scale (0 = normal to 6 = maximal impairment). The combined scores for the SKAMP are obtained by summing the values of all 13 items in the assessment. The range of SKAMP combined score is 0-78, with higher values represent a worse outcome.
Time Frame: Baseline to Day 15
Population: intent to treat population, placebo and dasotraline 4mg. The dasotraline 6mg arm was discontinued after 20 subjects were enrolled and no data were collected for this Arm/Group
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 51 | 52 | 0
Units on a scale | 1.99 (0.949) | -3.19 (0.942) |
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Least squares means, SEs, effect sizes, 95% CIs, and p-values were generated using an ANCOVA model, with treatment (dasotraline/placebo), mean SKAMP-CS at baseline, and site as fixed effects. The dasotraline 6 mg/day treatment arm was discontinued in Version 3.00 of the protocol; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -5.18, 95% CI 2-sided [-7.565 to -2.802], Standard Error of Mean 1.200

2. Secondary Outcome: Change From Baseline at Day 15 in Mean Swanson, Kotkin, Agler, M-Flynn, and Pelham Rating Scale (SKAMP)Attention Subscale Score Obtained From the 7 Assessments Collected Across the 12-hour Classroom Day (12 to 24 Hours Postdose)
Description: The Swanson, Kotkin, Agler, M-Flynn, Pelham Rating Scale (SKAMP) scale is a 13-item independent observer rating of subject impairment of classroom observed behaviors. Each item is rated on a 7-point impairment scale (0 = normal to 6 = maximal impairment). The Attention Subscale scores for the SKAMP are obtained by summing the values of Items 1-4 in the assessment. The range of SKAMP Attention Subscale score is 0-24, with higher values represent a worse outcome.
Time Frame: Baseline to Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 51 | 52 | 0
units on a scale | 0.79 (0.281) | -0.67 (0.279) |

3. Secondary Outcome: Change From Baseline at Day 15 in Mean Swanson, Kotkin, Agler, M-Flynn, and Pelham Rating Scale (SKAMP)-Deportment Subscale Score Obtained From the 7 Assessments Collected Across the 12-hour Classroom Day (12 to 24 Hours Postdose)
Description: The Swanson, Kotkin, Agler, M-Flynn, Pelham Rating Scale (SKAMP) scale is a 13-item independent observer rating of subject impairment of classroom observed behaviors. Each item is rated on a 7-point impairment scale (0 = normal to 6 = maximal impairment). The Deportment Subscale scores for the SKAMP are obtained by summing the values of Items 5-8 in the assessment. The range of SKAMP Deportment Subscale score is 0-24, with higher values represent a worse outcome.
Time Frame: Baseline to Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 51 | 52 | 0
units on a scale | 0.16 (0.356) | -1.44 (0.350) |

4. Secondary Outcome: Change From Baseline at Day 15 in Permanent Product Measure of Performance (PERMP)-Attempted and Correct Problems Scores Obtained From the 7 Assessments Collected Over the 12-hour Classroom Day (12-24-hours Postdose)
Description: TThe Permanent Product Measure of Performance (PERMP) is a math test consisting of 400 problems. Both attempted problems and correct problems are assessed. Subjects are to complete as many problems as possible in 10 minutes. Performance is measured by the number of math problems attempted and the number of math problems correctly completed. The minimum possible score is 0. The highest possible score is 400, with higher scores mean higher performance and less severe ADHD symptoms.
Time Frame: Baseline to Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 51 | 52 | 0
units on a scale
  attempted | -1.07 (5.871) | 22.60 (5.780) |
  corrected | -1.96 (5.864) | 22.09 (5.777) |
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Least squares means, SEs, effect sizes, 95% CIs, and p-values were generated using an ANCOVA model, with treatment (dasotraline/placebo), PERMP at baseline, and site as fixed effects. The dasotraline 6 mg/day treatment arm was discontinued in Version 3.00 of the protocol; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 23.67, 95% CI 2-sided [8.987 to 38.346], Standard Error of Mean 7.395
Statistical Analysis 2: Comparison: Placebo vs Dasotraline 4mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = 24.05, 95% CI 2-sided [9.381 to 38.714], Standard Error of Mean 7.389

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/56 | 0/20
Other Adverse Events (participants affected / at risk) | 14/56 | 24/56 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | Dasotraline 4mg (N=56) | Dasotraline 6mg (N=20)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | Dasotraline 4mg (N=56) | Dasotraline 6mg (N=20)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 4 (4)
Musle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 6 (6) | 1 (1)
Affect lability (Psychiatric disorders) | 4 (4) | 5 (5) | 4 (4)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Emotional poverty (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination tactile (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hallucination visual (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (8) | 5 (5)
Irritability (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish

DOCUMENTS (2):
  • Study Protocol (2017-09-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02734693/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT02734693/SAP_001.pdf